CLINICAL TRIAL: NCT02262533
Title: Drug Interaction Study of Apixaban and Atenolol in Healthy Subjects
Brief Title: Phase 1 Drug Interaction Study of Apixaban and Atenolol in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-033
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: N/A - Healthy Subjects
MeSH Terms: interventions — apixaban; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: Apixaban (Experimental): Apixaban tablet by mouth on specified day
  Interventions: Drug: Apixaban
- Treatment B: Atenolol (Experimental): Atenolol tablet by mouth on specified day
  Interventions: Drug: Atenolol
- Treatment C: Apixaban and Atenolol (Experimental): Apixaban and Atenolol tablets by mouth on specified day
  Interventions: Drug: Apixaban; Drug: Atenolol

INTERVENTIONS:
Drug: Apixaban
  Arms: Treatment A: Apixaban; Treatment C: Apixaban and Atenolol
Drug: Atenolol
  Arms: Treatment B: Atenolol; Treatment C: Apixaban and Atenolol

SUMMARY:
The purpose of this study is to assess the effect of Atenolol 100 mg on the Pharmacokinetics (PK) of Apixaban and the effect of Apixaban 10 mg on the PK of Atenolol in Healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECGs), and clinical laboratory determinations

Exclusion Criteria:

* Any significant acute or chronic medical illness, history of hypotension, history or evidence of abnormal bleeding or coagulation disorders, significant head injury within the last 2 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Apixaban and Atenolol plasma concentration | Days 1-13
  Blood samples for Atenolol PK were collected on days 1-3 of each period (Treatment B and C). Blood samples for Apixaban PK were collected on days 1-4 of each period (Treatment A and C)

SECONDARY OUTCOMES:
Safety and Tolerability based on adverse events (AE) reports and the results of vital sign measurements, electrocardiogram (ECGs), physical examinations, and clinical laboratory tests | Days 1-13

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bms Clinical Research Center, Hamilton, New Jersey, United States